CLINICAL TRIAL: NCT04419272
Title: Methylphenidate for the Treatment of Epilepsy-related Cognitive Deficits: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Methylphenidate for the Treatment of Epilepsy-related Cognitive Deficits
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA New York Harbor Healthcare System (U.S. Federal Agency); Portland VA Medical Center (U.S. Federal Agency); Miami VA Healthcare System (U.S. Federal Agency); VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NURD-003-22S; CX002474 (Other: eRA)
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
Keywords: attention; memory; cognition; seizure
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Methylphenidate; Lactose

STUDY DESIGN:
Intervention Model Description: Parallel group (methylphenidate vs. placebo), followed by open-label methylphenidate
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled study. A designated unblinded study team member will perform the randomization and provide group assignment to the local Research Pharmacies. The unblinded study team member and Research Pharmacies will hold the randomization key, while all other individuals are blinded to study group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Methylphenidate (Experimental): Subjects who will receive methylphenidate in the double-blinded period; when assigned to the active drug, the dosage of MPH will begin at 10mg twice per day, at 8am and 12pm, for one week. The dosage will then increase to 20mg twice daily, at 8am and 12pm, for the next 7 weeks.
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): Subjects who will receive placebo in the double-blinded period; when assigned to receive the placebo during the double-blinded period, subjects will be given a sugar pill for 8 weeks. The sugar pill will be taken twice per day, at 8am and 12pm.
  Interventions: Other: Placebo
- Open-Label Methylphenidate (Other): All subjects will be offered open-label methylphenidate during Weeks 9-16. the dosage of MPH will begin at 10mg twice per day, at 8am and 12pm, for one week. The dosage will then increase to 20mg twice daily, at 8am and 12pm, for the next 7 weeks.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — 10mg twice per day, at 8am and 12pm, for one week, then increased to 20mg twice daily, at 8am and 12pm, for the next 7 weeks during the double-blinded period.
  Other Names: Concerta, Ritalin, Daytrana, Aptensio XR, Metadate CD, Methylin, Quillivant XR, Jornay PM, Adhansia XR, Cotempla
  Arms: Methylphenidate
Other: Placebo — When assigned to receive the placebo during the double-blinded period, subjects will be given a sugar pill for 8 weeks. The sugar pill will be taken twice per day, at 8am and 12pm.
  Other Names: sugar pill, lactose
  Arms: Placebo
Drug: Methylphenidate — During the open-label extension phase, dosing will begin at 10mg twice per day, at 8am and 12pm, for one week. The dosage will then increase to 20mg twice daily, at 8am and 12pm, for the next 7 weeks.
  Other Names: Concerta, Ritalin, Daytrana, Aptensio XR, Metadate CD, Methylin, Quillivant XR, Jornay PM, Adhansia XR, Cotempla
  Arms: Open-Label Methylphenidate

SUMMARY:
Methylphenidate (MPH) is a stimulant, FDA-approved for the treatment of attention deficit hyperactivity disorder (ADHD). It is unknown, however, if stimulants would be of benefit for memory and thinking problems due to epilepsy. In this study, participants will be assigned randomly (i.e., by flip of a coin), to a group that takes MPH and a group that takes a placebo (sugar pill). Participants will not know the group to which they have been assigned. Tests of attention and memory will be completed before taking the study pills and at Week 8. All participants will then have the option of taking MPH for the next two months, and attention and memory will be tested again at Week 16. The study will determine whether methylphenidate is helpful for the treatment of attention and memory problems in adults with epilepsy, and whether the medication is safe and beneficial when taken over an extended time period.

DETAILED DESCRIPTION:
The proposed study is a randomized, double-blind trial of MPH vs. placebo in subjects with epilepsy and impaired attention. In the blinded phase, subjects will receive placebo or MPH (titrated to 20mg twice daily) for 8 weeks. Subjects will then receive open-label MPH for 8 weeks (titrated to 20mg twice daily). Cognitive tests will be performed at baseline, Week 8 (the end of the double-blind period), and at Week 16 (the end of the open-label period).

The primary aim is to evaluate the efficacy of MPH for the treatment of attentional dysfunction in subjects with epilepsy. It is expected that subjects will have improved attention when taking MPH compared to placebo, measured by the Conner's Continuous Performance Test (CPT). The effects of MPH on other cognitive functions that rely in part on attention, including a composite measure of memory (MCG Paragraph Test), psychomotor speed (Symbol Digit Modalities Test), and divided attention, psychomotor speed, and response inhibition (Stroop Color Word Interference Test), will be ascertained. Improved performance when taking MPH compared to placebo is expected. Finally, the study will establish the effect of MPH on overall quality of life. It is hypothesized that there will be improvement in self-reported quality of life with MPH, but no change with placebo, as assessed by the Quality of Life in Epilepsy Patient Inventory.

We will evaluate the safety of MPH compared to placebo with respect to seizure frequency. Secondary analyses will determine continued efficacy over an open-label period. To control for practice effects, cognitive performance will be compared to healthy subjects and epilepsy patients without cognitive complaints, who will complete the repeated cognitive measures but remain untreated for the duration of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. SUBJECTS WITH EPILEPSY

   Participants will include adult subjects with focal-onset epilepsy, based on clinical history, imaging studies and ictal and/or interictal EEG interpreted by a clinical epileptologist. Seizures may be symptomatic, idiopathic, traumatic, or non- traumatic in etiology. Subjects must have self-reported cognitive dysfunction. Subjects must also meet the following eligibility criteria:
   * Age 18 years of age or older;
   * Capacity to provide informed consent;
   * Ability to live independently and complete activities of daily living;
   * Stable seizure frequency at the time of enrollment, such that the subject's treating physician does not believe a change in ASM regimen to be warranted during the trial (ASMs should remain unchanged during the 16 weeks of participation unless absolutely required clinically due an unanticipated change in seizure frequency or severity);
   * Fluency in written and spoken English.
2. CONTROLS *DO NOT UNDERGO ANY DRUG OR PLACEBO INTERVENTION Two additional subject groups will be included, to control for effects of repeated testing in the open-label extension phase: healthy subjects and epilepsy patients without cognitive complaints, who will not receive the study drug at any point during the study. Epilepsy patients without cognitive deficits must otherwise meet all of the above criteria.

Healthy controls must meet the following inclusion criteria:

* Age 18 years or older;
* Capacity to provide informed consent;
* Ability to live independently and complete activities of daily living;
* Fluency in written and spoken English.

Exclusion Criteria:

SUBJECTS WITH EPILEPSY

Subjects with epilepsy with or without cognitive complaints will be excluded from participation for:

* Psychogenic, non-epileptic spells
* Delirium in the past year
* Other progressive neurologic illness (i.e., malignant brain tumor). A benign, stable neoplasm with no plans for resection will not be cause for exclusion.
* A history of alcohol or illicit drug abuse;
* Generalized tonic-clonic or other generalized motor seizure(s) within 48 hours or focal-onset seizures with impaired awareness within 24 hours of neuropsychological testing;
* Status epilepticus in the past year;
* Neurosurgery within the past 6 months;
* Suicide attempt in the past year and/or high-risk suicide flag in the medical record;
* Psychotic disorders
* Severe anxiety (>26 on the Beck Anxiety Inventory [BAI]) and impulse control disorders;
* Untreated sleep disorders;
* Use of narcotic or other sedating medications within 6 hours of testing (i.e., diphenhydramine);
* Concurrent severe major medical illness (i.e., cancer requiring chemotherapy or resection)
* Prior transient ischemic attack (TIA) or stroke

Subjects with epilepsy will also be excluded for a diagnosis of dementia (i.e., Alzheimer's disease). Subjects with epilepsy and cognitive complaints must have a MoCA score of 18 or greater. Subjects with epilepsy and no cognitive complaints must have a MoCA score of 26 or greater.

Subjects with epilepsy and cognitive complaints must meet additional exclusion criteria, to minimize risks of MPH:

* Current pregnancy or pregnancy planned during the trial
* Breastfeeding
* Concurrent treatment with a monoamine oxidase inhibitor (MAOI) or MAOI use within 14 days of beginning the trial;
* Structural cardiac abnormalities, cardiomyopathy, serious arrhythmias, or coronary artery disease (including a history of myocardial infarction, cardiac stent placement, coronary artery bypass graft surgery, or angina);
* Bipolar disorders;
* Concurrent use of medications for erectile dysfunction (e.g., tadalafil, sildenafil);
* Use of medications that may lower seizure threshold (e.g., tramadol, bupropion) or induce psychosis (i.e., varenicline);
* Known allergy or intolerance to MPH;
* Uncontrolled hypertension;

HEALTHY CONTROLS

Healthy controls will be excluded based on the following criteria:

* History of seizures, epilepsy, or psychogenic, non-epileptic spells;
* Diagnosis of dementia (i.e., Alzheimer's disease), MoCA score of <26;
* Delirium in the past year;
* Other progressive neurologic illness (i.e., malignant brain tumor);
* Prior moderate or severe traumatic brain injury (TBI);
* Mild TBI within the past 6 months;
* A history of alcohol or illicit drug abuse;
* Suicide attempt in the past year and/or high-risk suicide flag in the medical record;
* Psychotic, severe anxiety (BAI >26), or impulse control disorders;
* Untreated sleep disorders;
* Use of narcotic or other sedating medications within 6 hours of testing;
* Ongoing major neurological or medical illness (i.e., cancer requiring chemotherapy or resection);
* Prior TIA or stroke;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Conners Continuous Performance Test (CPT), Following Placebo vs. Methylphenidate | Week 8
  Conners Continuous Performance Test (CPT) d' value, a measure of attention, compared post-placebo vs. post-methylphenidate (MPH) in a double-blind, parallel group, placebo controlled, randomized design

SECONDARY OUTCOMES:
Change in Composite Measure of Cognition, Following Placebo vs. Methylphenidate | Week 8
  Scores on the MCG Paragraph (immediate and delayed recall), Symbol Digit Modality Test (SDMT), and Stroop tasks will be integrated into an omnibus outcome variable by combining performance based upon z-scores derived from normative tables. The omnibus score will be compared following placebo vs. active drug treatment.
Change in Overall Quality of Life, Following Placebo vs. Methylphenidate | Week 8
  Self-reported quality of life, as assessed by the Quality of Life in Epilepsy Inventory (QOLIE-89), compared post-placebo vs. post-methylphenidate. Range of scores 0-100, with higher scores representing better quality of life.
Change in Composite Measure of Cognition, Post-Open-Label | Week 16
  Scores on the MCG Paragraph (immediate and delayed recall), Symbol Digit Modality Test (SDMT), and Stroop tasks will be integrated into an omnibus outcome variable by combining performance based upon z-scores derived from normative tables. The omnibus score will be compared across baseline, Week 8, and post-open-label (Week 16)
Change in Subjective Cognitive Function, Following Placebo vs. Methylphenidate | Week 8
  Self-reported cognitive function, as assessed by the attention/concentration subscale of the Quality of Life in Epilepsy Inventory (QOLIE-89), compared post-placebo vs. post-methylphenidate.
Change in Subjective Cognitive Function, Post-Open-Label | Week 16
  Self-reported cognitive function, as assessed by the attention/concentration subscale of the Quality of Life in Epilepsy Inventory (QOLIE-89), compared across baseline, Week 8, and post-open-label (Week 16)
Change in Overall Subjective Quality of Life, Post-Open-Label | Week 16
  Self-reported quality of life, as assessed by the Quality of Life in Epilepsy Inventory (QOLIE-89), compared across baseline, Week 8, and post-open-label. Range of scores 0-100, with higher scores representing better quality of life.
Effects on Seizure Frequency | Week 8, Week 16
  Seizure occurrence will be recorded in a diary, with frequency compared across baseline, Week 8, and Week 16
Change in Conner's Continuous Performance Test (CPT), Post-Open-Label | Week 16
  Conners Continuous Performance Test (CPT) d' value, a measure of attention, with change compared across baseline, Week 8, and post-open-label (Week 16)
Change in Conners Continuous Performance Test (CPT), Comparing Methylphenidate Group to Untreated Controls | Week 8, Week 16
  CPT d' will be compared over the corresponding time periods in the methylphenidate, untreated epilepsy, and healthy control groups
Change in Digit Span Following Placebo vs. Methylphenidate | Week 8
  Total Digit Span score, compared post-placebo vs. post-methylphenidate. Range of scores 0-48, with higher scores indicating better performance.
Change in Digit Span, Post-Open-Label | Week 16
  Total Digit Span score, with change compared across baseline, Week 8, and post-open-label (Week 16)
Visual Paired Comparison Task Novelty Preference Score Following Placebo vs. Methylphenidate | Week 8
  Novelty preference score (range 0-100%), compared post-placebo vs. post-methylphenidate. Higher scores indicate better performance. (Manhattan site only)

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Leeman-Markowski, MD, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (4):
- United States (4):
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA NY Harbor Healthcare System, New York, NY, New York, New York
  - VA Portland Health Care System, Portland, OR, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
An anonymized data set may be shared upon written request to the PI and available no later than one year following publication. The data will be shared pending a written agreement 1) prohibiting the recipient from identification or re-identification of the data and forbidding any attempts to do so, and 2) allowing scientific use only. The data set will be provided via encrypted VA email.
Supporting Information: Study Protocol
Time Frame: Data will be made available no later than one year following publication. Data will be available for at least 6 years following completion of the study.
Access Criteria: The data will be shared pending a written agreement 1) prohibiting the recipient from identification or re-identification of the data and forbidding any attempts to do so, and 2) allowing scientific use only.